CLINICAL TRIAL: NCT06763068
Title: BIA-measured Skeletal Muscle Mass Used to Assess Frailty in Older Gastric Cancer Patients
Brief Title: Skeletal Muscle Mass Used to Assess Frailty in Older Gastric Cancer Patients
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yinning Guo, PhD student, Nanjing Medical University
Other Study IDs: 2020-273-2
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Gastric (Stomach) Cancer; Frailty; Sarcopenia; Malnutrition Elderly
Keywords: gastric cancer; skeletal muscle mass; frailty; sarcopenia
MeSH Terms: conditions — Stomach Neoplasms; Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Skeletal muscle mass and frailty — Measurement correlation variable

SUMMARY:
The primary aim of this study was to quantify the diagnosis of pre-surgical skeletal muscle mass in elderly gastric cancer patients and to analyse its correlation with frailty. The second aim was to investigate whether skeletal muscle mass, or sarcopenia, is associated with mobility and nutritional status, and anxiety and depression. The main questions it aims to answer are whether skeletal muscle mass is significantly associated with frailty and whether it can be used as a brief screening tool for preoperative frailty.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric cancer by endoscopy or pathology; age >60 years old; radical gastrectomy was proposed; be able to communicate simply in writing and verbal.

Exclusion Criteria:

* received preoperative radiotherapy or chemotherapy; combined with other sites of malignant tumors; combined with severe heart, liver, lung and renal insufficiency; recent using hormones, immunosuppressants; with physical disabilities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sampling method was used to select older people with gastric cancer who attended a tertiary care hospital in China from March 2021 to December 2022 as the study objects
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass | Within 24 hours of admission
  Skeletal muscle mass was measured by bioelectrical impedance analysis(BIA) and was classified as sarcopenia if it was less than 7.0 kg/m2 in men and 5.7 kg/m2 in women.
frailty | Within 24 hours of admission and discharge
  The Tilburg frailty scale was used to assess the frailty of older people with gastric cancer. The Tilburg frailty scale was compiled by Gobbens et al. The scale contains 15 items in three dimensions of physical, psychological and social frailty. The total score of the scale is 0-15 points and the cut-off value of the total scale was 5, with higher score indicating more severe frailty.

SECONDARY OUTCOMES:
Nutritional Status | Within 24 hours of admission and discharge
  The Mini Nutritional Assessment Short-form (MNA SF) scale was used to assess the nutritional status of older people with gastric cancer, which was a simplified version of the MNA scale developed by Rubenstein et al[. The total score of this scale is 14, 12~14 points indicate normal nutrition, 8~11 points indicate the risk of nutrition, ≤7 points indicate malnutrition.
anxiety and depression | Within 24 hours of admission and discharge
  Anxiety and Depression in older people with gastric cancer were assessed by the Chinese version of the Hospital Anxiety and Depression Scale (HADS), which was developed by Zigmond AS et al[23]. The scale has 14 items, 7 of which are used to assess depressed and 7 of which are used to assess anxiety. Each item has a score of 1-4 point and a total score of more than 7 indicates the presence of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The article has not yet been published